CLINICAL TRIAL: NCT02537314
Title: Role of the Foregut in Nutrient Metabolism in Lean and Obese Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Naji Abumrad, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 131032; R01DK100431 (NIH)
Record Dates: First submitted 2015-08-25; First posted 2015-09-01 (Estimated); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Obesity
Keywords: Normal Body Weight
MeSH Terms: conditions — Obesity | interventions — Benzocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- benzocaine (Active Comparator): 0.5% benzocaine solution in saline/hydrochloric acid administered by intraduodenal infusion one time (6 ml bolus followed by 75 ml/hour for 105 minutes)
  Interventions: Drug: benzocaine
- placebo (Placebo Comparator): Placebo (saline) solution administered by intraduodenal infusion one time (6 ml bolus followed by 75 ml/hour for 105 minutes)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: benzocaine — 0.5% benzocaine solution in saline/hydrochloric acid administered by intraduodenal infusion one time (6 ml bolus followed by 75 ml/hour for 105 minutes)
  Other Names: ethyl 4-aminobenzoate
  Arms: benzocaine
Other: placebo — Placebo (saline) solution administered by intraduodenal infusion one time (6 ml bolus followed by 75 ml/hour for 105 minutes)
  Other Names: NaCl, sodium chloride
  Arms: placebo

SUMMARY:
The overall hypothesis of this proposal is that nutrient sensing in the foregut regulates metabolic hormone secretion and nutrient metabolism via enteric neural signals, and these mechanisms might be defective in obesity.

DETAILED DESCRIPTION:
The study proposes two specific aims Aim 1 will determine if blocking enteric neuronal signaling will alter: a) circulating levels of nutrient substrates and secretion of hormones that regulate nutrient metabolism; and b) glucose and fatty acid absorption, production, and utilization.

Obese (BMI = 30-50 kg/m2) subjects will be studied. The topical anesthetic benzocaine will be infused into the duodenum prior to infusion of glucose and oleic acid into the duodenum. Duodenal infusions with a naso-intestinal feeding tube will circumvent the confounding effects of gastric emptying on the metabolic responses to a meal. Substrates (glucose, free fatty acids), and lipoproteins) and hormones will be measured by standard biochemical and immunological methods. Aim 2 will determine if enteric neural signals regulate appetite. The studies will be carried out in both lean and obese humans and the procedure will be performed as described above. In addition, the subjects will be asked to use a visual analog scale to estimate their level of appetite before, during and after enteral infusions.

ELIGIBILITY:
Inclusion Criteria:

* BMI 19 - 25 kg/m2 or 30 - 50 kg/m2
* Age 20 - 50 years

Exclusion Criteria:

* Contraindication to a nasoduodenal feeding tube (e.g., deviated nasal septum, prior upper gastrointestinal bleed, or history of easy bleeding)
* Prior gastric or intestinal surgery or pancreas resection
* Females with a positive pregnancy test
* Known history of intestinal diseases including, but not limited to, inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), celiac sprue
* Type 1 or type 2 diabetes
* Recent presence of or treatment for gastroenteritis (diarrhea and/or vomiting), constipation, or upper respiratory infection
* Anemia
* Abnormal electrocardiogram
* Prior adverse reaction to anesthesia
* Tobacco use

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-09; Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Hormones | 5 Hours
  Plasma levels of Cholecystokinin, gastric inhibitory peptide and glucagon like peptide and Ghrelin
Pancreatic Hormones | 5 Hours
  Plasma levels of Insulin, C-peptide, Glucagon
Glucose and Free Fatty Acids | 5 Hours
  Plasma levels

SECONDARY OUTCOMES:
Glucose Metabolism | 5 Hours
  Glucose tracer kinetics ([3-tritiated] glucose and [U-13C-carbon] oleate)
Fat Metabolism | 5 Hours
  Oleate tracer kinetics ([U-13 C-carbon] oleate)

OTHER OUTCOMES:
Appetite, Hunger, and GI symptoms | 5 Hours
  Visual Analog Scales (Likert)

CONTACTS AND LOCATIONS:
Overall Officials: Sinju Sundaresan, PhD, Principal Investigator — Vanderbilt University Medical Center; Naji N Abumrad, MD, Principal Investigator — Vanderbilt University Medical Center; Kala Dixon, MS, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Sundaresan S, Johnson C, Dixon KB, Dole M, Kilkelly D, Antoun J, Flynn CR, Abumrad NN, Tamboli R. Intraduodenal nutrient infusion differentially alters intestinal nutrient sensing, appetite, and satiety responses in lean and obese subjects. Am J Clin Nutr. 2023 Sep;118(3):646-656. doi: 10.1016/j.ajcnut.2023.06.011. Epub 2023 Aug 8. PMID 37661107